CLINICAL TRIAL: NCT01217619
Title: A Single Arm, One Center, Phase Ⅱ Study of Erlotinib as Neoadjuvent Treatment in Patients With Endobronchial Ultrasound Confirmed Stage ⅢA N2 NSCLC With EGFR Mutation in Exon 19 or 21
Brief Title: Erlotinib as Neoadjuvant Treatment in Patients With Stage ⅢA N2 NSCLC With Activating EGFR Mutation.
Acronym: ML25444
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baohui Han (Other)
Responsible Party: Sponsor-Investigator, Baohui Han, Vice President, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25444
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: neoadjuvant treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erlotinib (Experimental): Single-arm
  Interventions: Drug: erlotinib

INTERVENTIONS:
Drug: erlotinib — erlotinib 150mg/d continuously for 56 days
  Other Names: Tarceva

SUMMARY:
This is a single arm, one center, phaseⅡ study evaluating efficacy and safety of erlotinib as neoadjuvent treatment in patients with EBUS confirmed stage ⅢA N2 NSCLC with activating EGFR mutation in exon 19 or 21.

DETAILED DESCRIPTION:
Screening phase:

Patients clinically diagnosed as stage ⅢA N2 lung caner by CT technique will be pathologically proven as NSCLC with N2 by EBUS. The pathology specimen will be detected EGFR mutation by DNA sequencing. The patients with EGFR mutation in exon 19 or 21 will be enrolled in this study.

Neoadjuvant treatment phase:

Patient will receive erlotinib 150mg/day. Treatment will be scheduled to continue for a total of 8 weeks or disease progression or unacceptable toxicities.

Surgery treatment phase:

Tumor response will be evaluated with CT scan after 8 weeks of induction treatment. The patients with responsive disease considered to be technique resectable will undergo resection.

Post-surgery phase:

It is the discretion of the investigator whether the patient is a candidate for post-operative treatment which is considered to be in the best interest of the patients. It is recommended that patients with positive margins or residual tumor after surgery should receive radiation therapy. Patients after surgery will receive long-term follow-up including chest CT scan every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent provided. Males or females aged ≥18 years. Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.

Stage IIIA N2 NSCLC according to the pathological evidence of endobronchial ultrasound(EBUS).

The biopsy specimen shows EGFR mutation in exon 19 or 21 by DNA sequencing. Measurable disease must be characterized according to RECIST criteria: measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥20cm with conventional techniques (PE, CT, XR, MRI) or as ≥ 10cm with spiral scan.

ECOG performance status 0-1. Life expectancy ≥12 weeks.

Female subjects should not be pregnant or breast-feeding.

Exclusion Criteria:

The biopsy specimen shows EGFR wildtype in exon 19 or 21 by DNA sequencing. Patients with prior exposure to agents directed at the HER axis (e.g. erlotinib, gefitinib, cetuximab, trastuzumab).

Patients with prior chemotherapy or therapy with systemic anti-tumour therapy (e.g. monoclonal antibody therapy).

Known hypersensitivity to Tarceva or any of its recipients.

Evidence of any other disease, neurological or metabolic dysfunction, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the subject at high risk for treatment-related complications.

Sexually active males and females(of childbearing potential) unwilling to practice contraception during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-03-02 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
radical resection rate | operation after effective neoadjuvant treatment of tarceva for 56 days
  To evaluate radical resection rate of Tarceva as neoadjuvant treatment in patient with EBUS confirmed stage ⅢA N2 NSCLC with EGFR mutation in exon 19 or 21.

SECONDARY OUTCOMES:
Pathological Complete Remission | operation after effective neoadjuvant treatment of tarceva for 56 days
  To evaluate Pathological Complete Remission (pCR) rate of Tarceva as neoadjuvant treatment in patient with EBUS confirmed stage ⅢA N2 NSCLC with EGFR mutation in exon 19 or 21.
Objective Response Rate | Objective Response Rate measured by RECIST criteria in ITT population treated by erlotinib
  To evaluate Objective Response Rate (ORR) of Tarceva as neoadjuvant treatment in patient with EBUS confirmed stage ⅢA N2 NSCLC with EGFR mutation in exon 19 or 21.
disease free survival | From surgery to disease relapse or death
  To evaluate disease free survival(DFS) of Tarceva as neoadjuvant treatment in patient with EBUS confirmed stage ⅢA N2 NSCLC with EGFR mutation in exon 19 or 21.
overall survival | From study treatment to death due to any cause
  To evaluate overall survival(OS) of Tarceva as neoadjuvant treatment in patient with EBUS confirmed stage ⅢA N2 NSCLC with EGFR mutation in exon 19 or 21.
quality of life | During study treatment period
  To evaluate quality of life(QOL) of Tarceva as neoadjuvant treatment in patient with EBUS confirmed stage ⅢA N2 NSCLC with EGFR mutation in exon 19 or 21.
safety profile | For all the patient accepted study treatment
  To evaluate the safety profile using NCI CTC AE(version 4.0)
explorative biomarkers | During study conduction period
  To evalutate the relationship between biomarker and Tarceva neoadjuvent treatment efficacy (TBD).

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xiong L, Lou Y, Bai H, Li R, Xia J, Fang W, Zhang J, Han-Zhang H, Lizaso A, Li B, Gu A, Han B. Efficacy of erlotinib as neoadjuvant regimen in EGFR-mutant locally advanced non-small cell lung cancer patients. J Int Med Res. 2020 Apr;48(4):300060519887275. doi: 10.1177/0300060519887275. Epub 2019 Dec 29. PMID 31885349
- [Derived] Xiong L, Li R, Sun J, Lou Y, Zhang W, Bai H, Wang H, Shen J, Jing B, Shi C, Zhong H, Gu A, Jiang L, Shi J, Fang W, Zhao H, Zhang J, Wang J, Ye J, Han B. Erlotinib as Neoadjuvant Therapy in Stage IIIA (N2) EGFR Mutation-Positive Non-Small Cell Lung Cancer: A Prospective, Single-Arm, Phase II Study. Oncologist. 2019 Feb;24(2):157-e64. doi: 10.1634/theoncologist.2018-0120. Epub 2018 Aug 29. PMID 30158288